CLINICAL TRIAL: NCT05374785
Title: A 12-week, Phase II, Multicentre, Randomised, Double Blind, Efficacy and Safety Study Comparing CPL409116 to Placebo, in Combination With Methotrexate in Participants With Active Rheumatoid Arthritis Who Have an Inadequate Response to MTX
Brief Title: Efficacy and Safety Study Comparing CPL409116 to Placebo in Participants With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celon Pharma SA (Industry)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03JAK2021
Record Dates: First submitted 2022-05-04; First posted 2022-05-16 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; JAK inhibitors; Phase II
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: In all treatment arms the investigated product/ placebo is to be administered orally in a blinded fashion. In order to maintain the blind and minimize bias, all subjects will receive the same number and types of tablets each day of treatment (4 tablets BID)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CPL409116 60mg (Experimental): 60 mg BID of CPL409116
  Interventions: Drug: CPL409116
- CPL409116 120mg (Experimental): 120 mg BID of CPL409116
  Interventions: Drug: CPL409116
- CPL409116 240mg (Experimental): 240 mg BID of CPL409116
  Interventions: Drug: CPL409116
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CPL409116 — CPL409116 contained in the tablet called PG242 (60 mg)
  Arms: CPL409116 120mg; CPL409116 240mg; CPL409116 60mg
Other: Placebo — Tablets without CPL409116 as an active substance
  Arms: Placebo

SUMMARY:
The purpose of the following phase II clinical trial is to determine safety and effectiveness of Janus kinases and Rho-kinases inhibitor (JAK/ROCKi) in patients with Rheumatoid arthritis after oral administration of investigational medicinal product (IMP) called CPL409116. JAK inhibitors are a new class of small molecule drugs that modulate inflammatory pathways by blocking one or more JAK receptors. In recent years, JAK inhibitors have emerged as a new option for the treatment of various inflammatory diseases, including rheumatoid arthritis, psoriatic arthritis, skin disorders and others. CPL409116 inhibits JAK1 and JAK3 with less inhibitory activity against JAK2 and Tyk2. Inhibition of these kinases decreases inflammatory cytokine release which in turn decreases lymphocyte activation and proliferation. Moreover, CPL409116 blocks Rho-kinases (ROCKs), which are involved in diverse cellular processes including actin cytoskeleton organization, cell adhesion and motility, proliferation, apoptosis as well as smooth muscle contraction. ROCKs signalling is one of the major pathways implicated in the pathogenesis of cardiovascular, renal as well as fibrotic diseases. However recent data indicate their role in immune cell regulation and inflammatory disease development. CPL409116 was designed predominantly for the therapy of immune-related diseases: rheumatoid arthritis (RA) or psoriasis but the unique mode of action of this compound may be beneficial for patients suffering from fibrotic complications developing on the basis of autoimmune diseases. RA is a chronic systemic autoimmune disease characterised by persistent joint inflammation leading to loss of joint function as well as cartilage and bone damage. Chronic, progressive course of the disease results in disability, reduced quality of life, as well as higher comorbidity and mortality rates. It is well documented that JAK kinases play a pivotal role in cytokine receptor signalling to phosphorylate and activate signal transducer and activator of transcription (STAT) proteins. Several of these JAK-controlled cytokine receptor pathways are immediately involved in the initiation and progression of RA pathogenesis. After preclinical studies conducted by Celon Pharma, CPL409116 could have been classified as a good clinical candidate for the treatment of patients with RA and next, results obtained after the phase I clinical trial in healthy volunteers confirmed its safety and a good pharmacokinetic profile.

DETAILED DESCRIPTION:
This is to be a 12-week, phase II, multicentre, randomised, double blind, efficacy and safety study of CPL409116 in participants with active rheumatoid arthritis who are taking methotrexate but have an inadequate response to this drug. Eligible subjects are to be randomised into one of the 4 treatment arms (60 mg BID, 120 mg BID, 240 mg BID of CPL409116 or palcebo) and approximately 100 male and female subjects are to be enrolled in the study (25 patients per arm). The study is to include the screening period, the treatment period and the follow-up period. In all treatment arms the investigated product/ placebo is to be administered orally for 12 weeks in a blinded fashion. In order to maintain the blind and minimize bias, all subjects will receive the same number and types of tablets each day of treatment. In the screening period, patients are to undergo screening assessments from Day -28 to Day 0. Rolling admission is to be employed in this study. Patients that fulfil all the inclusion criteria and none of the exclusion criteria will be considered eligible for this study. During the treatment period, patients are to be dosed with 60, 120, 240 mg CPL409116 administered twice a day or placebo administered twice a day for 85 consecutive days (Day 1 to Day 85). The MTX dosage which should be orally or parenterally administered by participants during the study and before the start of the study should be in the range of 15-25 mg/ week, which is typical of current clinical practice. MTX must be applied for at least 12 weeks prior to Screening, and with no change in dosage and route of administration for at least 8 weeks prior to Day 1/ baseline. Within the follow-up period patients are to undergo safety assessment for 4 weeks after the last dose of IMP.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75 years at the time of signing informed consent;
2. Meets ACR/EULAR 2010 RA Classification Criteria with a duration of RA disease of ≥6 months at time of screening and participant not diagnosed before 16 years of age;
3. Must have active disease at both screening and baseline, as defined by having all three listed below:

   1. ≥ 6/68 tender/painful joints (TJC);
   2. ≥ 6/66 swollen joints (SJC);
   3. DAS28> 3,2.

   NOTE: If surgical treatment of a joint has been performed, that joint cannot be counted in the TJC or SJC for enrolment purposes.
4. Must have a C-reactive protein (CRP) measurement ≥7 mg/L at screening;
5. Must meet Class I, II or III of the ACR 1991 Revised Criteria for Global Functional Status in RA;
6. Must have inadequate response, despite currently taking Methotrexate (MTX): weekly 15-25 mg oral or injected (subcutaneous or intramuscular) for at least 12 weeks prior to Screening, and with no change in dosage and route of administration for at least 8 weeks prior to Day 1/ baseline. A lower dose of ≥10 mg/week is acceptable if reduced for reasons of side effects or intolerance to MTX, e.g. nausea/vomiting, hepatic or hematologic toxicity (there must be clear documentation in the medical record);
7. If using oral GCS must be on stable dose (equivalent to ≤10mg/day of prednisone) for at least 4 weeks prior to Day 1/ baseline;
8. If using NSAIDs must be on stable dose for at least 4 weeks prior to Day 1/ baseline;
9. A woman must be either:

   1. Not of childbearing potential:

      * postmenopausal (>45 years of age with amenorrhea for at least 12 months, without using exogenous hormonal contraception and with FSH ≥ 40 IU/L);
      * permanently sterile (hysterectomy, bilateral salpingectomy; bilateral oophorectomy); or otherwise be incapable of pregnancy.

      NOTE: premenopausal women who have had a bilateral tubal ligation/occlusion are considered capable of becoming pregnant.
   2. Of childbearing potential and using a double contraception including a barrier method (condom or occlusive cap) and a highly effective method of birth control (listed below):

   NOTE: highly effective methods of contraception are defined as:
   * established use (i.e. at least 8 weeks prior to Day 1) of combined (estrogen and progesterone) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal, injectable) or progesterone-only hormone contraception associated with inhibition of ovulation (oral, injectable);
   * intrauterine device (IUD) or intrauterine hormone-releasing system (IUS);
   * bilateral tubal occlusion/ligation;
   * vasectomized partner (vasectomized partner should be the sole partner for that subject and the absence of sperm should be confirmed).

   NOTE: sexual abstinence, defined as refraining from heterosexual intercourse throughout the study and for 12 weeks after the last IMP dose, is acceptable as a sole contraception method when this is in line with the preferred and usual lifestyle of the subject.
10. Participant (a man) who is sexually active with a woman of childbearing potential must agree to use a double contraception including a barrier method (male condom) and a highly effective method of contraception (highly effective method of contraception are listed above) during the study and 12 weeks after the last dose of CPL409116/ placebo administration.

    NOTE: Male subjects are responsible for informing his partner(s) of the risk of becoming pregnant and for reporting any pregnancy to the study doctor.

    NOTE: Participants (males and females) are furthermore willing to use contraception methods for 12 weeks after the last dose of CPL409116/ placebo administration. It is crucial to maintain appropriate methods of contraception if it is planned to continue methotrexate administration after the end of the study.
11. A woman of childbearing potential must have a negative blood pregnancy test (β -human chorionic gonadotropin [β-hCG]) at screening and negative urine pregnancy test on Day1/ baseline;
12. Informed Consent Form signed and dated prior to Screening evaluations;
13. Ability and willingness to comply with the requirements of the study Protocol;
14. Negative result of the COVID-19 RT-PCR test (real-time reverse transcription polymerase chain reaction) for the qualitative detection of nucleic acid coming from SARS- CoV-2 before inclusion to the study (Screening- 72 h before Day1/ baseline).

Exclusion Criteria:

1. Has had a serious infection (e.g. sepsis, pneumonia, pyelonephritis or any other serious infection as per Investigator's judgement), or has been hospitalized or received intravenous antibiotics for an infection within 3 months prior to Day 1/ baseline;
2. Any active infection including localized infections within 2 weeks prior to baseline;
3. History of opportunistic or recurrent (3 or more of the same infection requiring anti-infective treatment in any rolling 12-month period) infection;
4. History of chronic infections requiring anti-infective treatment within 6 months prior to Screening;
5. Subjects with a high risk of infection in the Investigator's opinion (e.g. subjects with leg ulcers, indwelling urinary catheter);
6. History of infected joint prosthesis or other implanted device with the retention of prosthesis or device in situ;
7. Symptomatic herpes zoster within 3 months prior to Screening;
8. History of disseminated herpes simplex infection or disseminated/complicated herpes zoster;
9. Hereditary or acquired immunodeficiency disorder, including immunoglobulin deficiency;
10. Known infection with human immunodeficiency virus (HIV) or positive test at Screening;
11. Presence of any of the following laboratory abnormalities at Screening:

    1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels ≥1.5 x the upper limit of normal (ULN);
    2. Absolute neutrophil count of <1.5 x 10^9/L (<1500/mm^3);
    3. Absolute lymphocyte count of <0.75 x 10^9/L (<750/mm^3);
    4. Absolute white blood cell (WBC) count of < 3.0 x 10^9 /L (<3000/mm^3);
    5. Hemoglobin <9.0 g/dL (90 g/L);
    6. Thrombocytopenia, as defined by a platelet count <100 x 10^9/L (< 100 000/mm^3) at Screening;
    7. Total bilirubin ≥1.5× the upper limit of normal (ULN).
12. Current or history of clinically significant (per Investigator's judgment) liver or biliary disease or significantly abnormal liver function test at screening (ALT or AST level ≥ 1.5 x ULN and/or total bilirubin ≥1,5× the upper limit of normal (ULN);
13. Current acute or chronic HCV and/or HBV infection:

    1. Subjects who are seropositive for antibodies to hepatitis C virus (at Screening) may be allowed to participate in the study provided they have 2 negative HCV RNA test results 6 months apart after completing antiviral treatment and prior to Screening, and have a third negative HCV RNA test result at Screening.
    2. HBV serology:

       * a positive result for HBsAg will be exclusionary;
       * a positive result for anti-HBc antibodies in subjects negative for HBsAg requires HBV DNA testing. A positive test result for HBV DNA will be exclusionary;
       * For subjects who are negative for HBsAg and anti-HBc antibodies and has had a HBV vaccination a positive test result for anti-HBs antibodies is expected - such subjects may be enrolled without HBV DNA testing. In non-vaccinated patients positive for anti-HBs antibodies HBV DNA testing is required;
       * a positive result for HBV DNA will be exclusionary.

    NOTE: enrolled subjects positive for anti-HBc antibodies and/or anti-HBs antibodies (except for vaccinated subjects negative for anti-HBc antibodies and positive for anti-HBs antibodies) will have repeated HBV DNA testing at week 6 (or early termination visit) and last follow-up visit. A positive result for HBV DNA testing in these subjects will require immediate interruption of study drug and a hepatologist consultation.
14. Current or history of clinically significant renal disease (per investigation judgment) or eGFR<60mL/min/1.73m^2;
15. Breast cancer or other malignancy (including lymphoma, leukemia) within the past 5 years except for cervical carcinoma in situ that has been completely resected with no evidence of recurrence or metastatic disease for at least 12 months or cured basal cell carcinoma with no evidence of recurrence for at least 12 months;
16. History of major organ transplant (e.g. kidney, heart, liver, lung) or hematopoietic stem cell/bone marrow transplant;
17. History of lymphoproliferative disease or signs/ symptoms suggestive of possible lymphoproliferative disease, including splenomegaly of lymphadenopathy;
18. History or current moderate to severe congestive heart failure (New York Heart Association [NYHA] class III or IV), or within the last 6 months, a cerebrovascular accident, myocardial infarction, unstable angina, unstable arrhythmia or any other cardiovascular condition which, in the opinion of the investigator, would put the subject at risk by participation in the study;
19. History or presence of other significant concomitant illness that, according to the Investigator's judgment, would place the participant at unacceptable risk when taking investigational product or could interfere with the interpretation of data;
20. History of other (than RA) chronic inflammatory arthritis or systemic autoimmune disorder other than Sjögren's syndrome secondary to RA, that may confound the evaluation of the effect of the study intervention such as mixed connective tissue disease, psoriatic arthritis, juvenile chronic arthritis, spondyloarthritis, Felty's Syndrome, systemic lupus erythematosus, scleroderma, Crohn's disease, ulcerative colitis, or vasculitis;
21. Presence of fibromyalgia that, in the Investigator's opinion, would make it difficult to appropriately assess RA activity for the purposes of this study;
22. Undergone any major surgery within 8 weeks prior to study entry or will require major surgery during the study that, in the opinion of the Investigator would pose an unacceptable risk to the participant;
23. Current or previous active Mycobacterium tuberculosis (TB) regardless of treatment;
24. Evidence of latent TB (as documented by a positive QuantiFERON-TB test at Screening, no findings on medical history or clinical examination consistent with active TB, and a normal chest radiograph);
25. Previous household contact with a person with active tuberculosis (TB) and did not receive appropriate and documented prophylaxis for TB;
26. Clinically significant multiple or severe drug allergies or severe post-treatment hypersensitivity reactions (including, but not limited to erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis);
27. Inherited or acquired thrombophilia and/ or current or history of thromboembolic events/ disease;
28. Screening 12-lead ECG that demonstrates relevant abnormalities that, in the opinion of the Investigator, are clinically significant and indicate an unacceptable risk for the subject's participation in the study (eg, QTc >450 msec or a QRS interval >120 msec). If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the subject's eligibility;
29. Pregnancy or breast- feeding.

    NOTE: Women of childbearing potential must have a negative pregnancy test at Screening, at randomization and at scheduled visits throughout the study.
30. Narcotic and alcohol addiction or abuse (more than 14 alcohol units per week: one unit = 150 mL wine, 360 mL beer, 45 mL 40 % spirits) (UK guidelines);
31. Positive drug screen or alcohol breath tests;
32. Blood donation within the last month before Day1/ baseline;
33. Current therapy with any disease-modifying antirheumatic drugs (DMARDs) other than MTX. All DMARDs (except for MTX) must be ceased before Day 1/ baseline, as follows:

    * 1 month before: etanercept, sulfasalazine, chloroquine/ hydroksychloroquine;
    * 3 months before: leflunomide (4 weeks in case of cholestyramine washout);
    * 3 months before: adalimumab, golimumab, infliksimab, certolizumab, tocilizumab, gold, cyclosporine, penicillamine, azathioprine.
34. Previous use of (at any time):

    1. cyclophosphamide
    2. tacrolimus
35. Previous use of JAK inhibitors;
36. Previous use of biologic agent other than tocilizumab or TNF-alpha inhibitor. Previous use of one (and only one) biologic agent (tocilizumab or TNF-alpha inhibitor) is allowed if administered for less than 3 months or ceased because of other than lack of effectiveness causes;
37. Vaccinated with a live vaccine (i.e. containing live or attenuated pathogens) within 3 months before Day 1/ baseline or necessity to vaccinate during the clinical trial.

NOTE: Investigators should ensure that all study enrolment criteria have been met at Screening and on Day 1. If a patient status after Screening changes at baseline (Day 1) such that the study patient no longer meets all eligibility criteria, then the patient should be excluded from participation in the study (such patient is to be considered as screen failure). History or presence of any other medical or psychiatric condition, or laboratory abnormality that, in the opinion of the Investigator, may place the subject at unacceptable risk for study participation or may interfere with the study results should be considered as an exclusion criterion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Change in Disease Activity Score 28 joint count C reactive protein (DAS28(CRP)). | Baseline to Week 12
  Change from baseline in Disease Activity Score 28 joint count C reactive protein (DAS28(CRP)) score at Week 12
  DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28- (CRP) will be calculated from swollen joint count (SJC) and tender/painful joint count (TJC) using 28 joints count, CRP [mg/L] and patient global assessment of disease activity on a 100 millimeter (mm) visual analog scale (VAS: scores ranging from 0 mm [very well] to 100 mm [extremely bad], higher scores indicate worse health condition).
  Score interpretation:
  <2.6 suggests disease remission. 2.6-3.2 suggests low disease activity >3.2-5.1 suggests moderate disease activity >5.1 suggest high disease activity

SECONDARY OUTCOMES:
Proportion of patients with remission over time assessed by Disease Activity Score 28 joint count C reactive protein (DAS28(CRP)). | Baseline through Week 12
  Proportion of patients with Disease Activity Score 28 joint count C reactive protein (DAS28(CRP)). score< 2.6
  DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28- (CRP) will be calculated from swollen joint count (SJC) and tender/painful joint count (TJC) using 28 joints count, CRP [mg/L] and patient global assessment of disease activity on a 100 millimeter (mm) visual analog scale (VAS: scores ranging from 0 mm [very well] to 100 mm [extremely bad], higher scores indicate worse health condition).
  Score interpretation:
  <2.6 suggests disease remission. 2.6-3.2 suggests low disease activity >3.2-5.1 suggests moderate disease activity >5.1 suggest high disease activity
Proportion of patients achieving American College of Rheumatology (ACR) ACR20/50/70/90 response over time | Baseline through Week 12
  Proportion of patients achieving American College of Rheumatology (ACR) ACR20/50/70/90 response over time.
  The specific components of the ACR Assessments (ACR Core Dataset) that are to be used in this study are:
  1. Tender/Painful Joint count (TJC) (68);
  2. Swollen Joint Count (SJC) (66);
  3. Patient's Assessment of Arthritis Pain;
  4. Patient's Global Assessment of Arthritis;
  5. Physician's Global Assessment of Arthritis;
  6. C-Reactive Protein (CRP);
  7. Erythrocyte Sedimentation Rate (ESR);
  8. Health Assessment Questionnaire - Disability Index (HAQ-DI).
  Participants with 20/50/70 and 90% improvement in 68-tender and 66-swollen joint counts and 20/50/70 and 90% improvement respectively in at least 3 of the 5 measures: patient's global assessment of arthritis, physician global assessment of arthritis, patient's assessment of arthritis pain, health assessment questionnaire-disability index(HAQ-DI) and CRP.
Change in the Tender/Painful and Swollen Joint Count | Baseline through Week 12
  Change from baseline in the Tender/Painful and Swollen Joint Count
  Sixty-eight (68) joints will be assessed to determine the number of joints that are considered tender or painful. The response to pressure/motion on each joint will be assessed using the following scale: Present/Absent/Not Done/Not Applicable- artificial joints will not be assessed.
Change in the Physician's Global Assessment (PhGA) of Arthritis | Baseline through Week 12
  Change from baseline in the Physician's Global Assessment (PhGA) of Arthritis
  The investigator will assess how the patient's overall arthritis appears at the time of the visit. This is an evaluation based on the patient's disease signs, functional capacity and physical examination, and should be independent of the Patient's Global Assessment of Arthritis. The investigator's response will be recorded using a 100 mm visual analogue scale (VAS).
  VAS measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Incidence and severity of adverse events, serious adverse events, and withdrawals due to adverse events | Baseline through Week 16
  Incidence and severity of adverse events, serious adverse events, and withdrawals due to adverse events
Incidence of abnormality in clinical chemistry parameters | Baseline through Week 16
  Incidence of abnormality in clinical chemistry parameters
Incidence of abnormality in hematological parameters | Baseline through Week 16
  Incidence of abnormality in hematological parameters
Change in blood pressure measurement | Baseline through Week 16
  Change from baseline in blood pressure measurement
  Number of Participants with Change in blood pressure measurement
Change in pulse rate measurement | Baseline through Week 16
  Change from baseline in pulse rate
  Number of Participants with Change in pulse rate measurements
Change in temperature measurement | Baseline through Week 16
  Change from baseline in temperature
  Number of Participants with Change in temperature measurements
Change in the Patient's Assessment of Arthritis Pain (PAAP;visual analogue scale [VAS] | Baseline through Week 12
  Change from baseline in the Patient's Assessment of Arthritis Pain (PAAP) visual analogue scale (VAS)
  Patients will assess the severity of their arthritis pain using a 100 mm visual analogue scale (VAS) by placing a mark on the scale between 0 (no pain) and 100 (most severe pain), which corresponds to the magnitude of their pain.
Change in the Patient Global Assessment of Arthritis (PtGA, VAS-visual analogue scale ) | Baseline through Week 12
  Change from baseline in the Patient Global Assessment of Arthritis (PtGA, visual analogue scale, VAS)
  Patients will answer the following question, "Considering all the ways in which your rheumatoid arthritis affected you, how do you feel about your arthritis today?" VAS measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Change from baseline in the Health Assessment Questionnaire - Disability Index (HAQ-DI) | Baseline through Week 12
  HAQ-DI evaluate the degree of difficulty a participant has experienced during the past week in 8 categories of daily living activities: dressing/grooming; arising; eating; walking; reach; grip; hygiene; and other activities over past week.
  Scoring is from 0 (without any difficulty) to 3 (unable to do).
Change in the Short Form Survey (SF-36 RAND) | Baseline to Week 12
  Change from baseline in the Short Form Survey (SF-36 RAND) 8 domain scores and physical component score (PCS) and mental component score (MCS).
  Short Form Survey (SF-36 RAND) is a 36-item generic health status measure.
Change in the Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) total score | Baseline to Week 12
  Change from baseline in the Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) total score.
  The FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week.Instrument scoring yields a range from 0 to 52, with higher scores representing better patient status (less fatigue).
CPL409116 and metabolite M3 pharmacokinetic variable: AUC(0-6h) | up to 6 hours after administration of IMP on Day 1, 8, 57 and 85
  Pharmacokinetic Endpoint: area under the plasma concentration - time curve from time 0 to 6 hours after IMP administration
CPL409116 and metabolite M3 pharmacokinetic variable: Cmax | up to 6 hours after IMP administration on Day 1, 8, 57 and up to 24 hours after IMP administration on Day 85
  Pharmacokinetic Endpoint: The maximum concentration of the CPL409116 compound in plasma after IMP administration, obtained directly from the measured concentrations
CPL409116 and metabolite M3 pharmacokinetic variable: Tmax | up to 6 hours after administration of IMP on Day 1, 8, 57 andand up to 24 hours after IMP administration on Day 85
  Pharmacokinetic Endpoint: The time to reach the maximum plasma concentration (Cmax), obtained directly from the actual sampling times
CPL409116 and metabolite M3 pharmacokinetic variable: T1/2 (if possible) | up to 6 hours after IMP administration on Day 1, 8, 57 and up to 24 hours after IMP administration on Day 85
  Pharmacokinetic Endpoint: The plasma elimination half-life
CPL409116 and metabolite M3 pharmacokinetic variable: Kel (if possible) | up to 6 hours after IMP administration on Day 1, 8, 57 and up to 24 hours after IMP administration on Day 85
  Pharmacokinetic Endpoint: Kel is to be estimated via linear regression of time versus log of concentration
CPL409116 pharmacokinetic variables: C0 and C2.5h | 5 minutes before IMP administration and up to 2.5 hours after IMP administration on Day 29
  Pharmacokinetic Endpoint: the concentration pre-dose and 2.5 hours after IMP administration.

OTHER OUTCOMES:
MFI (median fluorescence intensity) or percentage of phosphorylated proteins | on Day 1; 29; 57 and 85
  CPL409116 ability to inhibit STAT and MYPT, MLC phosphorylation by inhibition of JAK and ROCK kinases activity in patients with active RA.

CONTACTS AND LOCATIONS:
Locations (10):
- Poland (7):
  - MICS Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Centrum Nowoczesnych Terapii Sp. z o.o. "Dobry Lekarz", Krakow
  - AMICARE Centrum Medyczne Sp. z o. o., Spółka Komandytowa, Lodz
  - Medyczne Centrum Hetmańska, Poznan
  - Samodzielny Publiczny Zespół Opieki Zdrowotnej w Tomaszowie Lubelskim, Tomaszów Lubelski
  - Wojskowy Instytut Medyczny, Warsaw
  - PCS Sp. z o. o., Łady
- Ukraine (3):
  - Medical center of the limited liability company "Medical center "Consilium Medical", Kyiv
  - Polyclinic of the center of medical services and rehabilitation JSC "Company of aviation and rocket technology manufacture", Kyiv
  - Communal enterprise "Hospital No. 1" of the Zhytomyr City Council, consulting and treatment department "Research Center", Zhytomyr

REFERENCES:
- [Derived] Wieczorek M, Kisiel B, Wlodarczyk D, Leszczynski P, Kurylchyk IV, Vyshnyvetskyy I, Kierzkowska I, Pankiewicz P, Kaza M, Banach M, Kogut J. Dual JAK and ROCK inhibition with CPL'116 in patients with rheumatoid arthritis with inadequate response to methotrexate: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Rheumatol. 2025 Sep;7(9):e629-e641. doi: 10.1016/S2665-9913(25)00060-8. Epub 2025 Jun 11. PMID 40516565

DOCUMENTS (2):
  • Study Protocol (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT05374785/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/85/NCT05374785/SAP_001.pdf